CLINICAL TRIAL: NCT04189185
Title: Suture Fixation Versus Tension Band Wiring of Simple Displaced Olecranon Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aalborg University Hospital (Other)
Collaborators: Regionshospitalet Horsens (Other); Aarhus University Hospital (Other); Regionshospitalet Viborg, Skive (Other); Kolding Sygehus (Other); Randers Regional Hospital (Other)
Responsible Party: Principal Investigator, Andreas Haubjerg Qvist, MD, Principal investigator, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20190039
Record Dates: First submitted 2019-11-19; First posted 2019-12-06 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: Olecranon Fracture
MeSH Terms: conditions — Olecranon Fracture

STUDY DESIGN:
Intervention Model Description: Two study arms. One arm is treated with k-wire tension band wiring and one leg is treated with suture fixation
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: An envelope deciding the treatment modality is drawn while the patient is anesthetized. Post operative follow-up is performed by blinded assessors. The treatment will be revealed after one year, or if the patient is excluded from the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- K-wire tension band wiring (Active Comparator): The patient is treated with 1.6 mm k-wires and 1 mm cerclage
  Interventions: Procedure: Suture fixation
- Suture fixation (Active Comparator): The fracture is reduced and fixed with 2.0 Orthocord suture.
  Interventions: Procedure: Suture fixation

INTERVENTIONS:
Procedure: Suture fixation — The fracture is reduced. A 2.5 mm hole is drilled in the dorsal olecranon 15mm from the fracture. A suture is passed through the hole and is fixed to the triceps muscle. A second suture is fixed to the triceps muscle in a figure 8 configuration.

SUMMARY:
Simple displaced olecranon fractures are most often treated with tension band wiring. This is an effective treatment, but the risk of subsequent re-operation is high. The investigators propose open reduction and internal fixation with a strong suture, thus reducing the risk of re-operation significantly.

DETAILED DESCRIPTION:
Background Olecranon fractures are frequent with an incidence of 11.5 per 100.000 people per year. Olecranon fractures are classified according to the Mayo classification in three groups. Type 1A and B are treated conservatively, while comminute fractures of type Mayo 2B and 3B are treated with plate osteosynthesis.

The most common type is a simple two part fracture, Mayo type 2A, which represents 74% of all olecranon fractures. The typical treatment of Mayo type 2A fractures is osteosynthesis using k-wires and tension band wiring. This provides adequate fracture healing and good functional results. The use of plate osteosynthesis for Mayo type 2A fractures does not provide functional or health economic benefits compared with operation with tension band wiring.

Common for both techniques is a high risk of re-operation due to delayed healing of the surgical wound, and complications arising from the implanted material.

Recently, new techniques for Mayo type 2A fractures have been described, in which no metal is implanted. Osteosynthesis is achieved with strong sutures. These techniques have been shown to reduce the high risk of complications leading to re-operation without effecting the functional outcome or fracture healing rate.

Hypothesis The investigators hypothesize that suture fixation of Mayo type 2A fractures will decrease the risk of re-operation and provide equal functional outcome compared with tension band wiring.

Design Prospective, randomized multicenter study

ELIGIBILITY:
Inclusion Criteria:

* Olecranon fracture, Mayo Type 2A

Exclusion Criteria:

* Bilateral upper extremity fracture
* Open fracture
* Neurovascular affection
* Injury to ligament, dislocation or subluxation
* Additional upper extremity fracture
* Pathological fracture
* Previous elbow issue
* Fracture more than 14 days old
* Substance abuse
* medical contraindication for surgery
* Previous fracture to the same elbow

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2019-12-05 (Estimated); Primary Completion 2021-11-20 (Estimated); Study Completion 2023-11-20 (Estimated)

PRIMARY OUTCOMES:
Re-operation | 1 year
  The rate of re-operation

SECONDARY OUTCOMES:
The Disabilities of the Arm, Shoulder and Hand (DASH) Score | 1 year
  Patient reported outcome measure. Range from 0 (No disability) to 100 (most severe disability).
European Quality of life - 5 Dimensions (EQ-5D) questionnaire | 1 year
  Patient reported outcome measure. Score from 1 (best) to 3 (worst) in 5 different categories.
Range of motion | 1 year
  Range of motion in elbow
Sick days | 1 year
  Number of sick days/Return to work
Non-union | 6 months
  Rate of non-union
Rate of complications | 1 year
  Rate of complications to the treatment: Infection, nerve damage, delayed wound healing.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Qvist, MD, Principal Investigator — Aalborg University Hostipital; Andreas Haubjerg Qvist, MD, Principal Investigator — Aalborg University Hospital
Locations (1):
- Aalborg Sygehus - Farsø, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Duckworth AD, Clement ND, Aitken SA, Court-Brown CM, McQueen MM. The epidemiology of fractures of the proximal ulna. Injury. 2012 Mar;43(3):343-6. doi: 10.1016/j.injury.2011.10.017. Epub 2011 Nov 9. PMID 22077988
- [Background] Ates Y, Atlihan D, Yildirim H. Current concepts in the treatment of fractures of the radial head, the olecranon and the coronoid. J Bone Joint Surg Am. 1996 Jun;78(6):969. No abstract available. PMID 8666617
- [Background] Matar HE, Ali AA, Buckley S, Garlick NI, Atkinson HD. Surgical interventions for treating fractures of the olecranon in adults. Cochrane Database Syst Rev. 2014 Nov 26;2014(11):CD010144. doi: 10.1002/14651858.CD010144.pub2. PMID 25426876
- [Background] Duckworth AD, Clement ND, White TO, Court-Brown CM, McQueen MM. Plate Versus Tension-Band Wire Fixation for Olecranon Fractures: A Prospective Randomized Trial. J Bone Joint Surg Am. 2017 Aug 2;99(15):1261-1273. doi: 10.2106/JBJS.16.00773. PMID 28763412
- [Background] Helm RH, Hornby R, Miller SW. The complications of surgical treatment of displaced fractures of the olecranon. Injury. 1987 Jan;18(1):48-50. doi: 10.1016/0020-1383(87)90386-x. PMID 3440616
- [Background] Romero JM, Miran A, Jensen CH. Complications and re-operation rate after tension-band wiring of olecranon fractures. J Orthop Sci. 2000;5(4):318-20. doi: 10.1007/s007760070036. PMID 10982677
- [Background] Snoddy MC, Lang MF, An TJ, Mitchell PM, Grantham WJ, Hooe BS, Kay HF, Bhatia R, Thakore RV, Evans JM, Obremskey WT, Sethi MK. Olecranon fractures: factors influencing re-operation. Int Orthop. 2014 Aug;38(8):1711-6. doi: 10.1007/s00264-014-2378-y. Epub 2014 Jun 4. PMID 24893946
- [Background] Macko D, Szabo RM. Complications of tension-band wiring of olecranon fractures. J Bone Joint Surg Am. 1985 Dec;67(9):1396-401. PMID 3908460
- [Background] Phadnis J, Watts AC. Tension band suture fixation for olecranon fractures. Shoulder Elbow. 2017 Oct;9(4):299-303. doi: 10.1177/1758573216687305. Epub 2017 Jan 18. PMID 28932288
- [Background] Das AK, Jariwala A, Watts AC. Suture Repair of Simple Transverse Olecranon Fractures and Chevron Olecranon Osteotomy. Tech Hand Up Extrem Surg. 2016 Mar;20(1):1-5. doi: 10.1097/BTH.0000000000000106. PMID 26630656
- [Background] Nimura A, Nakagawa T, Wakabayashi Y, Sekiya I, Okawa A, Muneta T. Repair of olecranon fractures using fiberWire without metallic implants: report of two cases. J Orthop Surg Res. 2010 Oct 12;5:73. doi: 10.1186/1749-799X-5-73. PMID 20937160
- [Background] Hudak PL, Amadio PC, Bombardier C. Development of an upper extremity outcome measure: the DASH (disabilities of the arm, shoulder and hand) [corrected]. The Upper Extremity Collaborative Group (UECG). Am J Ind Med. 1996 Jun;29(6):602-8. doi: 10.1002/(SICI)1097-0274(199606)29:63.0.CO;2-L. PMID 8773720
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Gummesson C, Atroshi I, Ekdahl C. The disabilities of the arm, shoulder and hand (DASH) outcome questionnaire: longitudinal construct validity and measuring self-rated health change after surgery. BMC Musculoskelet Disord. 2003 Jun 16;4:11. doi: 10.1186/1471-2474-4-11. Epub 2003 Jun 16. PMID 12809562
- [Background] Hunsaker FG, Cioffi DA, Amadio PC, Wright JG, Caughlin B. The American academy of orthopaedic surgeons outcomes instruments: normative values from the general population. J Bone Joint Surg Am. 2002 Feb;84(2):208-15. doi: 10.2106/00004623-200202000-00007. PMID 11861726
- [Derived] Qvist AH, Christensen BB. Suture fixation versus tension band wiring in simple displaced olecranon fractures - a study protocol. Dan Med J. 2024 Oct 18;71(11):A01240038. doi: 10.61409/A01240038. PMID 39575943